CLINICAL TRIAL: NCT02065934
Title: Clinical Audit of Cardio Pulmonary Resuscitation Management in Adults Patient Units of Care by in Situ Simulation
Acronym: SIMACRIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Yannick BRUNIN, MD, Centre Hospitalier Universitaire de Besancon
Other Study IDs: EI/2013/116
Record Dates: First submitted 2014-01-13; First posted 2014-02-19 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: in Hospital Cardiac Arrest; in Situ Simulation; Clinical Audit; Education
Keywords: in hospital cardiac arrest; in situ simulation; clinical audit; education
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cardio-pulmonary resuscitation

SUMMARY:
Clinical audit of in-hospital cardiac arrest management by in situ simulation

Objectives: correct latent safety threats, knowledge gap, and crisis resource management (CRM)

Design: clinical audit, observational sudy. Primary outcome: In Hospital resuscitation scale. Exploratory outcomes: non technical skills, validated stress inventory, and questionnaire on perceptions of the simulation and organisational changes needed.

ELIGIBILITY:
Inclusion Criteria:

* team members: nurses, auxiliary nurses, residents, doctors, students

Exclusion Criteria:

* non volunteers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Team members
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
In-Hospital resuscitation scale | 5 months

SECONDARY OUTCOMES:
ANTS scale | 5 months
Peritraumatic Dissociative Experiences Questionnaire (PDEQ) | 5 months
  validated stress inventory
Peritraumatic Distress Inventory (PDI) | 5 months
  validated stress inventory

CONTACTS AND LOCATIONS:
Overall Officials: Yannick BRUNIN, Dr, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France